CLINICAL TRIAL: NCT05914584
Title: "Baricitinib for Treating Hospital-acquired Pneumonia in Critically Ill Patients With a Proinflammatory Phenotype, an International Phase II/Phase III, Randomized, Controlled Trial - TREAT-HAP Study.
Brief Title: "Baricitinib for Treating Hospital-acquired Pneumonia in Critically Ill Patients With a Proinflammatory Phenotype.
Acronym: TREAT-HAP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC22_0522
Record Dates: First submitted 2023-04-19; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Hospital-acquired Pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia | interventions — baricitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baricitinib + Standard of care (Experimental): Baricitinib injected per os for 10 days (4mg/day). the first administration of this treatment is performed within the 6 hours following the randomization, followed by daily administration for a total of 10 days.
  The standard of care : for treating HAP will comply with international guidelines. For all patients, empiri antimicrobial therapy is initiated imedialty after collecting the respiratory sample and can thus be started before the randomization to avoid delayed antimicrobial therapy. Its recommanded to broaden the spectrum in case of resistant bacteria resistant to the empirical antimicrobial therapy but il is not recommanded to prolong the antibiotic tratment for more than 7-8 days
  Interventions: Drug: Baricitinib 4 MG
- Standard of care alone (Sham Comparator): Same as described in arm 1
  Interventions: Drug: Baricitinib 4 MG

INTERVENTIONS:
Drug: Baricitinib 4 MG — Reference drug

SUMMARY:
The goal of this clinical trial is to determine the safety (phase II), then efficacy (phase III) of baricitinib plus standard of care (SOC) as compared to SOC alone for the treatment of hospital-acquired pneumonia in patients with a pro-inflammatory profile.

DETAILED DESCRIPTION:
For both groups :

At inclusion visit :

* Verification of inclusion and non-inclusion criteria
* Patient information and signature of consent form
* Pregnancy test (urine ou blood)
* Randomization
* Clinical evaluation (cardiac frequency, saturation, tracheal secretions, PaO2/FiO2 ratio, body temperature, mechanical ventilation support)
* Collection of respiratory fluid and blood for biobank
* Liver function test (AST, ALT, bilirubin), blood white cells count and EKG
* Treatment compliance
* Concomitant medications (antimicrobial therapy and steriods)
* Survival and EQ-5D-5L

At visit 1 to visit 10 ( Day1- day10)

* Clinical evaluation (cardiac frequency, saturation, tracheal secretions, PaO2/FiO2 ratio, body temperature, mechanical ventilation support)
* Study drug administration (daily)
* Collection of respiratory fluid and blood for biobank (day 3 and day 7)
* Liver function test (AST, ALT, bilirubin), blood white cells count and EKG (Liver, day 3 and day 7)
* Treatment compliance
* Adverse event
* Concomitant medications (antimicrobial therapy and steriods)

At visit 11(Day 10-12 test-of-cure) :

* Clinical evaluation (cardiac frequency, saturation, tracheal secretions, PaO2/FiO2 ratio, body temperature, mechanical ventilation support)
* Collection of respiratory fluid and blood for biobank
* Collection of the respiratory fluid for bacterial cure
* Liver function test (AST, ALT, bilirubin), blood white cells count and EKG
* Adverse event
* Concomitant medications (antimicrobial therapy and steriods)

At visit 12 :

* Adverse event
* Survival and EQ-5D-5L

At visit 13 (month 3) and visit 14 (month 6) :

* Query in NHI Database (SNDS) for consumption of Health resources (pharmaceuticals, consultations...)
* Survival and EQ-5D-5L
* Health -related quality of the life (SF-36), anxiety/depression (HADS), subjective well-being (SWLS)
* Interview with a researcher in pshychology (20 patients and their relatives - only in France)

ELIGIBILITY:
Inclusion Criteria:

* Ventilators-associated pneumonia (VAP) or hospital -acquired pneumonia requiring invasive ventilation (V-HAP)
* Diagnosis of HAP according to European guidelines : association of two clinical criteria (body temperature > 38°c and purulent pulmonary secretions), the appearance of a new infiltrate or change in an existing infiltrate on chest radography, and respiratory sample (AET, BAL, mini-BAL or blind BAL) collected for bacteriological diagnosis (results can be pending at inclusion). The diagnosis of HAP can have been made outside of ICU
* VAP : patients should have received machenical ventilation via an endotracheal or nasotracheal tube for the least 48h at the time of HAP diagnosis. V-HAP : patients should have been hospitalized for the least 48 hours before the onset of the first signs or symptoms and required invasive mechanical ventilation during HAP treatment
* Biological systemic inflammatory response defined according to the on-site standard of acre (CPR > 125 mg/L and/or PCT > 2µg/L and/or ferritin blood level > 650 ng/mL
* Receiving antimicrobal therapy for the current episode of HAP pneumonia for less than 72 hours
* Informed consent from legal representative or emergency procedure (when possible according to national regulation). If it's impossible to obtain patient consent before the inclusion (comatose patients), patient consent for the study continuation will be obtained as soon as deemed possible
* Person insured under a helth insurance scheme

Exclusion Criteria:

* Pregnant women (serum or urine test), breastfeeding woment
* Patient under legal protection (inc. under guardianship or trusteesheep)
* Hypersensitivity to baricitinib
* Uncontrolled herpes zoster, viral hepatitis, infection with human immunodeficiency virus, fungal infections or tuberculosis
* Severe hepatic insufficiency (child-Pugh B or C)
* Acute or chronic renal insufficiency (modification of diet in renal disease (MDRD) creatinine clearance < 30 ml/min/1.73 m²)
* Persistent anemia (haemoglobin < 8 g/L), lymphopenia (absolute lymphocyte < 500 cells/mm3)
* Immunosuppression (hematologic cancer, aplasia, chemotherapy/radiotherapy for cancer within 3 months prior to the inclusion or anti-graft rejection drug)
* Recent (<90 days) trhomboembolic event (venous trhombosis, pulmonary embolism, myocardial infarction, and/or stroke)
* Participation to an interventional drug study within 1 month prior to the inclusion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the safety (phase II), of baricitinib plus standard of care (SOC) as compared to (SOC) alone for the treatment of hospital-acquired pneumonia in patients with a pro-inflammatory profile | Day 28
  Using a hierarchic procedure. We will test the baricitinib superiority on the clinical cure rate at the test-of-cure visit realized 10-12 days after randomization or at the ICU discharge. If the superiority criterion is met at the test-of-cure visit, we will test the baricitinib superiority on the rate of all-cause mortality on Day 28
Determine the efficacy (phase III) of baricitinib plus standard of care (SOC) as compared to (SOC) alone for the treatment of hospital-acquired pneumonia in patients with a pro-inflammatory profile | Day 28
  Using a hierarchic procedure. We will test the baricitinib superiority on the clinical cure rate at the test-of-cure visit realized 10-12 days after randomization or at the ICU discharge. If the superiority criterion is met at the test-of-cure visit, we will test the baricitinib superiority on the rate of all-cause mortality on Day 28

SECONDARY OUTCOMES:
To demonstrate the efficacy of baricitinib on pneumonia-associated morbidity reduction | Day 28
  In case of a non-significant difference in the rate of clinical cure, the co-primary outcome will be presented as a secondary outcome.
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality reduction | Day 28
  In case of a non-significant difference in the rate of clinical cure, the co-primary outcome will be presented as a secondary outcome.
To demonstrate the efficacy of baricitinib on pneumonia-associated morbidity | Month 3 and Month 6
  All-cause morbidity at Month 3 and Month 6
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality | Month 3 and Month 6
  All-cause mortality at Month 3 and Month 6
To demonstrate the efficacy of baricitinib on pneumonia-associated morbidity reduction | Day 28
  Rate of pleural empyema at Day 28.
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality reduction | Day 28
  Presence of pleural empyema at Day 28.
To demonstrate the efficacy of baricitinib on pneumonia-associated morbidity reduction | Day 28
  Rate of microbial failure (defined as a positive respiratory culture at the ToC visit)
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality reduction | Day 28
  Rate of microbial failure (defined a a positive respiratory culture at the ToC visit)
To demonstrate the efficacy of baricitinib on pneumonia-associated morbidity reduction | Up to 28 days
  Rate of pneumonia relapse (defined as a second episode of HAP with one r more identical pathogens, rate of pneumonia recurrence (defined as a second epsode of AP with different pathogens)
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality reduction | Up to 28 days
  Rate of pneumonia relapse
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality reduction | Up to Day 28
  Time course of body temperature
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality reduction | Up to Day 28
  Cardiac pulse rate
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality reduction | Up to Day 28
  Oxygen saturation
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality reduction | Up to Day 28
  Type of mechanical ventilation support (invasive, noninvasive, none) (daily evaluation at 8.00am and 8.00pm)
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality reduction | Up to Day 12
  Leukocyte counts (every 48 hours) for 12 days
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality reduction | Day 28
  Pa02/FiO2
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality reduction | Day 28
  Rates of non respiratory hospital-acquired infections
To demonstrate the efficacy of baricitinib on pneumonia-associated morbidity reduction | Day 28
  Rates of nonrespiratory hospital-acquired infections
To demonstrate the efficacy of baricitinib on pneumonia-associated morbidity reduction | Day 28
  Antibiotic-free days (the number of antibiotic-free days is defined as the number of days between Day 1 and Day 28 for which living patients do not receive antibiotics.
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality reduction | Day 28
  Antibiotic-free days (the number of antibiotic-free days is defined as the number of days between Day 1 and Day 28). Dead patients will be ascribed 0 antibiotic-free days.
To demonstrate the efficacy of baricitinib on pneumonia-associated morbidity reduction | Up to Month 3
  Duration of invasive mechanical ventilation and invasive mechanical ventilation-free days (defined as the number of days between Day 1 and Month 3 for which living patients breath spontaneously.
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality reduction | Up to Month 3
  Duration of invasive mechanical ventilation and invasive mechanical ventilation-free days (defined as the number of days between Day 1 and Month 3). Dead patients will be ascribed 0 mechanical ventilation-free days.
To demonstrate the efficacy of baricitinib on pneumonia-associated mortality reduction | Up to Month 3
  Duration ogf hospitalization and hospital-free days (the number of hospital-free days is defined as the number of days between Day 1 and Month 3 which living patients are outside of a hospital.
To demonstrate the efficacy of baricitinib on pneumonia-associated morbidity reduction | Up to Month 3
  Duration ogf hospitalization and hospital-free days (the number of hospital-free days is defined as the number of days between Day 1 and Month 3). Dead patients will be ascribed 0 hospital-fre days)

OTHER OUTCOMES:
Determine the safety of baricitinib | Day 10-12
  Rate of serious adverse effects and suspected unexpected serious adverse reaction (SUSAR) at Day 28.
  Rate of neutropenia, lymphopenia and trhombocytosis at the test-of-cure visit (Day 10-12).
  Rates of drug-induced liver injury defined by the International DILI Expert Working Groups as ALT greater than or equal to 5 or ALP greater than or equal to 2 and TBL inferior to 2 ULN (corresponding to grade 1, mild severity) Rate of acute kidney failure (KDIO 2-3) at the test-of-cure visit (Day 10-12) Rate of major trhombo-embolic events at the test-of-cure visit (Days 10-12), rate of EKG modification at the test-of-cure visit (Day10-12)
Determine if baricitinib increases the economic efficiency of the treatment of pneumonia | 6 months
  Cost-effictiveness analysis (CEA) using QALYs (Quality-Adjusted Life-Years) will consist in estmating an incremental cost-effectiveness ratio (ICER)
Determine the suitability of baricitinib from the patient's perspectives | Up to 6 months
  Changes in health-related quality of life after randomization measured with the Short Form-36 scale validated in French, Spanish, Flemish and Dutch. These questionnaires will be filled in by the patient (patient's perspective) or by one relative if the patient cannot respond for him/herself (patient's perspective).
Determine the suitability of baricitinib from the patient's perspectives | Up to 6 months
  Changes in anxiety and depression measured with the Hospital and Aanxiety Depression scale validated in French, Spanish, Flemish and Dutch. These questionnaires will be filled in by the patient (patient's perspective) or by one relative if the patient cannot respond for him/herself (patient's perspective).
Determine the suitability of baricitinib from the patient's perspectives | Up to 6 months
  Changes in subjective well-being measured with the Satisfaction With Life Scale (SWLS) validated in French, Spanish, Flemish and Dutch.
To identify biomarkers for stratidication of patents into responders and non-responders to baricitinib | Day 10-12
  To capture the complexity of the host-pathogens interactions and to clinically validate biomarkers for the stratification of patients into low/high risk of poor outcomes of HAP and responders/non responders to immunotherapy
To identify a biobank of blood and respiratory samples collected from humans with hospital-acquired pneumonia | Day 10-12
  Collection of respiratory fluid and blood for biobank
Determine the safety of baricitinib | Day 28
  Rate of serious adverse effects and suspected unexpected serious adverse reaction (SUSAR) at Day 28.
Determine the safety of baricitinib | Day 10-12
  Rate of neutropenia, lymphopenia and thrombocytosis at the test-of-cure visit
Determine the safety of baricitinib | Day 10-12
  Rates of drug-induced liver injury defined by the International DILI Expert Working Groups as ALT greater than or equal to 5 or ALP greater than or equal to 2 and TBL inferior to 2 ULN (corresponding to grade 1, mild severity)
Determine the safety of baricitinib | Day 10-12
  Rate of acute kidney failure (KDIO 2-3) at the test-of-cure visit
Determine the safety of baricitinib | Day 10-12
  Rate of major thrombo-embolic events at the test-of-cure visit
Determine the safety of baricitinib | Day 10-12
  Rate of EKG modification at the test-of-cure visit

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ROQUILLY, Principal Investigator — Nantes University Hospital
Locations (24):
- Belgium (5):
  - St-Luc Clinics, Brussels
  - Ghent University Hospital, Ghent
  - Groupe Jolimont, Haine-Saint-Paul
  - Clinique Saint-Pierre, Ottignies
  - University Hospital of UCL Namur, Yvoir
- France (15):
  - CHU Angers, Angers
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CH La Roche sur Yon, La Roche-sur-Yon
  - CHU de Limoges, Limoges
  - CHU de Marseille, Marseille
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Beaujon, Paris
  - CHU la Pitié-Salpétrière, Paris
  - CHU Pitié-Salpétrière, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes
- University Medical Center Utrecht, Utrecht, Netherlands
- Spain (3):
  - Hospital Clinic, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided